CLINICAL TRIAL: NCT00074620
Title: A Randomised, Multicenter, Open-Label, Parallel Group Study to Assess the Safety of PEG-Hirudin (SPP200) Compared to Unfractionated Heparin as Anticoagulant Treatment in Patients Undergoing Haemodialysis Via an Arteriovenous Graft
Brief Title: A Clinical Study to Assess the Safety of PEG-Hirudin (SPP200) Compared to Heparin in Patients Who Are on Haemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Speedel Pharma Ltd. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPP200CRD01
Record Dates: First submitted 2003-12-17; First posted 2003-12-19 (Estimated); Last update posted 2007-10-05 (Estimated); Status verified 2007-10

CONDITIONS: Chronic Kidney Failure; Vascular Graft Occlusion
Keywords: Haemodialysis; PEG-Hirudin; Vascular graft occlusion; Renal replacement therapy; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Graft Occlusion, Vascular | interventions — polyethyleneglycol-hirudin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PEG-hirudin

SUMMARY:
The study will look at the safety profile (unwanted effects) of the long-lasting anticoagulant PEG-hirudin (SPP200) and compare these unwanted effects to those of unfractionated heparin, commonly used in haemodialysis to avoid clotting of the graft and of the haemodialysis machine.

ELIGIBILITY:
* Patients undergoing chronic haemodialysis via an arteriovenous graft
* Arteriovenous graft in place for at least 3 months
* Duration of haemodialysis of at least 3 months, with 3 full dialysis sessions per week with a duration between 2 and 5 hours per session
* Women patients must be either postmenopausal for more than 1 year or, if of childbearing age, must use adequate contraception
* Women patients must have a negative serum pregnancy test within one week of randomisation
* Able to provide written informed consent prior to study participation

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260
Dates: Start 2003-11; Study Completion 2006-01

PRIMARY OUTCOMES:
To determine the safety and tolerability of SPP200 in patients undergoing chronic haemodialysis via an arteriovenous graft.

SECONDARY OUTCOMES:
To determine the efficacy of PEG-hirudin compared to unfractionated heparin (UFH) on the frequency of vascular graft occlusions and on time to first graft occlusions.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M Mann, MD, PhD, Study Chair — Speedel Bio Ltd
Locations (1):
- Pennsylvania Hospital - Franklin Dialysis Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: The National Kidney Foundation is a voluntary organisation which seeks to prevent kidney diseases, improve the health of patients and increase the availability of organs for transplantation — http://www.kidney.org/
- See also: The American Association of Kidney Patients helps kidney patients and their families deal with the physical, emotional and social impact of kidney diseases — http://www.aakp.org/